CLINICAL TRIAL: NCT06679920
Title: IDEAL Phase II Study of a Newly Designed Optical Coherence Tomography Probe During Transurethral Resection for Optimizing Bladder Cancer Diagnosis and Treatment
Brief Title: Study With a Newly Optical Coherence Tomography Probe for Optimizing Bladder Cancer Diagnosis and Treatment
Acronym: BLOCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC (Other)
Responsible Party: Principal Investigator, Harrie P. Beerlage, Prof. dr. H.P. Beerlage, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL83449.018.23; ESTAR21207 (Other Grant/Funding Number: EUROSTARS)
Record Dates: First submitted 2024-11-05; First posted 2024-11-08 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Bladder Cancer
Keywords: OCT; Optical Coherence Tomography; Bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Optical coherence tomography measurements during transurethral resection of a bladder tumour (Other): Single arm
  Interventions: Device: Optical coherence tomography

INTERVENTIONS:
Device: Optical coherence tomography — Measurement with opctical coherence tomography of tumour and normal bladder tissue during transurethral resection of a bladder tumour (TURBT)

SUMMARY:
The goal of this clinical trial is to see if a new designed optical coherence tomography catheter can be used in bladder cancer in patients undergoing a transurethral resection of a bladder tumour. The main question it aims to answer is:

- Is the optical coherence tomography catheter feasible in capturing images of bladder tumours and normal bladder wall during a transurethral resection of a bladder tumour?

Participants will undergo measurements with a new optical coherence tomography device during the transurethral resection of their bladder tumour(s).

DETAILED DESCRIPTION:
Rationale:

Bladder cancer is the 10th most common form of cancer in the world with 573.278 new cases of bladder cancer and 212,536 deaths in 2020. Despite current treatment options, 5-year recurrence rates up to 78% have been reported. Therefore, frequent and long-term follow-up of bladder cancer patients is required. Up until now, the gold standard for diagnosing bladder cancer is cystoscopy with subsequent transurethral resection of the bladder tumour (TURBT). In certain cases a repeat-TURBT (re-TURBT) is necessary to ensure radicality and to confirm the stage of the tumour. The frequent cystoscopies and multiple operations result in a substantial burden for bladder cancer patients and in substantial healthcare costs. Therefore, finding other options to determine the tumour grading and staging by a so called 'optical biopsy' is necessary. This would enable other treatment options, such as out-patient laser fulguration or active surveillance reducing the subsequent TURBT after cystoscopy.

Optical coherence tomography (OCT) is an optical technique that uses infrared light to create high resolution, real-live images of tissue. OCT has been studied in the upper urogenital tract for urothelial carcinoma with good results. However, this is a different situation, since the ureter is a tubular structure with limited space and the tested OCT probe is a sideward looking probe. Previously, two different, forward looking, OCT probes have been studied in the bladder. The studies show different results on sensitivity and specificity. Some results are very promising, while others show no advantage for OCT over white light cystoscopy (WLC). However, the studied probes have a low frames per second (FPS) rate. This results in stammering images and makes the probes very sensitive for motion artefacts. Furthermore, both OCT catheters are not on the market (anymore). Since the OCT techniques have improved over the last decade, a new forward looking OCT probe has been developed. The newly designed OCT catheter has a much higher FPS rate and has used techniques to improve the resolution of the images. Therefore, the newly designed micro-electro-mechanical system (MEMS) based OCT catheter looks promising to improve the diagnosis and treatment of bladder cancer. The present study is an IDEAL stage-IIa feasibility study.

Objectives:

The primary objective:

- To investigate the feasibility of capturing in-vivo cross section images of the bladder wall in bladder cancer patients with the MEMS based OCT catheter.

Secondary objectives:

* To evaluate the duration of the OCT measurements.
* To determine the depth of invasion of the tumour based on OCT images and test if there is an association with the histopathological results of the resected tissue(s).
* To determine the grade of the tumour based on OCT images and test if there is an association with the histopathological results of the resected tissue(s).
* To determine if the OCT catheter is able to acquire evaluable images of resection beds.
* To compare the tumour grade and invasion estimated by the urologist during WLC with the tumour grade and invasion determined by the OCT images.

Study design: A prospective, mono-center, IDEAL stage IIa clinical study to investigate the feasibility of a newly designed MEMS based OCT catheter.

Study population: Patients that are >18 years old, who are electively planned for a TURBT are eligible for the study. A maximum of 25 will be included patients but inclusion is earlier completed when 15 technically successful ("feasible") procedures are performed.

Intervention: In the operation theatre, the urologist will introduce a rigid resectoscope and will perform a white light cystoscopy which are part of the standard procedure. The urologist will estimate the tumour invasion and tumour grade for each tumour. Then the OCT catheter is inserted through this rigid resectoscope which is used for the planned TURBT. Cross-sectional OCT images of the tumour(s) will be acquired as well as OCT images of one part of normal looking bladder wall contralateral to the tumour(s). A maximum of 5 tumours in each participant with a maximum diameter of 2 centimeter will be analysed with the OCT catheter. After the images are recorded, the TURBT will be performed. In case of multiple tumours, the resected tissue of the different tumours will be collected separately. After the TURBT is completed, the OCT catheter will be introduced again through the resectoscope to capture images of the resection bed(s). The resected tumour tissue will be send to the pathology laboratory as part of the standard procedure.

Main study parameters/endpoints:

The primary outcomes of this study are:

* Assessment of procedural feasibility of OCT measurement:

  o Procedural feasibility will be determined by the ability to generate images of the normal bladder wall and bladder tumour(s), as assessed by the operating urologist. Feasibility will be achieved if diagnostic images of the tumour and normal bladder are obtained in over 60% of the patients. Our aim is to obtain diagnostic images from 15 procedures, limiting the inclusion to a maximum of 25 patients.
* Analysis of feasibility based on image utilization:

  * Feasibility will also be assessed by determining the percentage of images suitable for diagnosis out of the total number obtained. A percentage exceeding 80% will be deemed feasible.

The secondary outcomes:

* The duration of the OCT measurements in minutes.
* The overall concordance between the OCT catheter diagnosis of tumour invasion (stage) compared with the pathological results of the resected tissue(s).
* The overall concordance between the OCT catheter diagnosis of tumour grade compared with the pathological results of the resected tissue(s).
* The ability of the OCT catheter to acquire evaluable images of the resection bed.
* The concordance between tumour grade and invasion estimated by the urologist during WLC and the tumour grade and invasion determined by the OCT images and histopathology.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: There is little burden for the patients. The only burden is a prolonged operation time which is expected to be approximately 20 minutes. It is assumed that there is hardly no additional risk for the patient, since the OCT catheter is inserted through the working channel of the resectoscope that is used for the TURBT The probe is designed with rounded corners. Additionally, the probe is not purposeful in contact with the bladder wall, since the focus point is approximately 1cm from the tip of the probe. Therefore, the risk of bladder perforation is not expected to be increased.

The probe is tested in vitro (use through the working channel of operating instruments, sterilization process is tested and according to GCP). Because the catheter is not tested in vivo, there is a very small chance of unexpected events related to the material, e.g. breaking of material, fragment loss inside bladder that can be removed by surgical instruments through the working channel.

There is no benefit for participants of this study. The burden and risks of this study are the same for all participants. The patients will receive the standard of clinical care during participation and the histopathological evaluation will not be affected by the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Have at least 1 suspected bladder tumour seen at cystoscopy.
* Have a bladder that is accessible for cystoscopy.
* Be in a physical condition to undergo a TURBT.
* Eligible patients must be fully informed about the study and written signed informed consent must be obtained prior to any study related investigation/intervention.

Exclusion Criteria:

* Pregnant or lactating women.
* The only tumour site is at the bladder neck.
* The tumour(s) is larger than 2 centimetres in diameter.
* >5 tumours present.
* Solely a suspected flat lesion present.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Procedural feasibility | During the TURBT
  The ability to generate images of the normal bladder wall and bladder tumour(s). Feasibility will be achieved if diagnostic images of the tumour and normal bladder are obtained in over 60% of the patients.
Image utilization feasibility | During the TURBT
  Feasibility will also be assessed by determining the percentage of images suitable for diagnosis out of the total number obtained. A percentage exceeding 80% will be deemed feasible.

SECONDARY OUTCOMES:
Duration of the measurements | During the TURBT
  The duration of the OCT measurements in minutes
Concordance tumour stage based on OCT with histopathology | From TURBT to histopathology result (approximately 4 weeks)
  The overall concordance between the OCT catheter diagnosis of tumour invasion (stage) compared with the pathological results of the resected tissue(s)
Concordance between tumour grade based on OCT and histopathology | From TURBT to histopathology result (approximately 4 weeks)
  The overall concordance between the OCT catheter diagnosis of tumour grade compared with the pathological results of the resected tissue(s).
Evaluable resection bed OCT images | During the TURBT
  The ability of the OCT catheter to acquire evaluable images of the resection bed.
Concordance OCT and WLC tumour stage and grade | From TURBT to histopathology result (approximately 4 weeks)
  The concordance between tumour grade and invasion estimated by the urologist during WLC and the tumour grade and invasion determined by the OCT images and histopathology.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Amsterdam University Medical Center, Amsterdam, North Holland
  - Amsterdam University Medical Center, Amsterdam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Remmelink MJ, Nieuwenhuijzen JA, de Bruin DM, Oddens JR. Newly Designed Optical Coherence Tomography Catheter for Optimizing Bladder Cancer Diagnosis and Treatment: Protocol for a Feasibility Study. JMIR Res Protoc. 2025 Dec 2;14:e76644. doi: 10.2196/76644. PMID 41329952